CLINICAL TRIAL: NCT01842282
Title: Clinical Protocol to Investigate the Efficacy of Amlexanox for Treatment of Glucose and Lipid Abnormalities in Obese Type 2 Diabetics
Brief Title: Amlexanox for Type 2 Diabetes and Obesity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to limited funding, trial was suspended, intending to restart with additional funds; then preliminary results were obtained, and research moved on to placebo controlled trial. Results for both have been published.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elif Oral, Professor of Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00065177
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Results first posted 2024-01-17 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus Type 2; Non Alcoholic Fatty Liver Disease; Obesity
Keywords: diabetes mellitus type 2; non alcoholic fatty liver disease; obesity; amlexanox
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Obesity | interventions — amlexanox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Amlexanox (Experimental)
  Interventions: Drug: Amlexanox

INTERVENTIONS:
Drug: Amlexanox
  Other Names: Solfa tablets

SUMMARY:
This study involves the use of a research drug, Amlexanox, for the treatment of type 2 diabetes, insulin resistance, obesity and non-alcoholic fatty liver disease (NAFLD). Amlexanox is taken orally in a pill three times a day. The investigators plan to continue therapy for a period of 12 weeks followed by a follow-up 4 weeks after therapy ends. The investigators will evaluate the changes in metabolic parameters (e.g. blood cholesterol, liver function, insulin resistance) and body composition characteristics (e.g. the pattern of fat distribution in the body). Seven eligible subjects in this study will also be evaluated for a change in liver disease by a liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old at baseline and <60 years of age.
* Is male, female not of childbearing potential, or meets all the following criteria if female of childbearing potential (including perimenopausal women who have had a menstrual period within one year):

  * Not breastfeeding.
  * Negative pregnancy test result (human chorionic gonadotropin, beta subunit [βhCG]) at baseline (not applicable to hysterectomized females).
  * Must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate when use consistently and correctly, such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire duration of study period.
* Has physician-confirmed diabetes mellitus with a clear diagnosis or per ADA criteria with fasting glucose>126 mg/dL or HbA1c >6.4% or 2 hour GTT >200 mg/dL or or pre-diabetes with fasting glucose >100 mg/dL (n= up to 8)
* BMI ≥27 and <36 kg/m2.
* On no medications or only on first line oral medications (such as Metformin and/or DPP IV inhibitors) for treatment of type 2 diabetes mellitus with a stable regimen for >12 weeks.
* Alcohol consumption of less than 40 grams/week.
* A liver US confirming presence of fatty infiltration of the liver.
* Is able to read, understand and sign the U of M IRBMED approved informed consent form (ICF), communicate with study physician and study team, understand and comply with protocol requirements.

Exclusion Criteria:

* On insulin, sulfonylurea or other injectables for treatment of type 2 diabetes
* Unable to conduct home based glucose monitoring
* HbA1c>9.5%
* Presence of advanced liver disease (as evidenced by abnormal synthetic function, abnormal PT or albumin).
* Evidence of other etiologies of viral hepatitis.
* Presence of hematologic, bone marrow and/or other abnormalities.
* Presence of hemoglobinopathy or other hematological abnormalities that will interfere with accurate measurement of HbA1c
* Presence of HIV infection.
* Inability to give informed consent.
* Presence of ESRD, any type of active cancer, or >class 2 congestive heart failure (New York Heart Association Functional Classification System), based on medical history and physical examination.
* Active chronic infection such as known chronic osteomyelitis or tb, etc. (may be transient).
* Creatinine >1.5 mg/dL
* Proliferative diabetic retinopathy, nonproliferative retinopathy is allowed
* Unable to ambulate
* Clinically relevant CAD: history of stent, CABG or cardiologist confirmed angina
* Any other condition in the opinion of the investigators that may impede successful data collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07-19 (Actual); Primary Completion 2014-02-25 (Actual); Study Completion 2014-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elif A Oral, MD, Principal Investigator — Univeristy of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Amlexanox: Amlexanox
Period: Overall Study
Arm/Group | Amlexanox
Started | 7
Completed | 6
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Amlexanox
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 60 [50 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
A1C [Mean (Full Range); unit: percent of total hemoglobin] | 7.9 [6.7 to 9.4]
Weight [Mean (Full Range); unit: kg] | 97.6 [83.1 to 122.7]
Hepatic Steatosis by MRI [Mean (Full Range); unit: percentage of fat in liver] | 7.5 [4.2 to 9.7]

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Change in HbA1c from baseline to 12 weeks as shown by mean increase or decrease of HbA1c where decreased values represent better health
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: percentage of total hemoglobin
Arm/Group | Amlexanox
Number analyzed (Participants) | 6
percentage of total hemoglobin | 0 [-0.6 to 0.6]

2. Primary Outcome: Hepatic Steatosis by MRI
Description: change in hepatic steatosis from baseline to 12 weeks: MRI Liver fat percentage as shown by mean difference
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: percentage of liver mass
Arm/Group | Amlexanox
Number analyzed (Participants) | 6
percentage of liver mass | -2.2 [-5.9 to 0.3]

3. Secondary Outcome: Weight
Description: Change in weight (Kg) from baseline to 12 weeks as shown by mean difference, where lower weights represent healthier outcomes
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: kg
Arm/Group | Amlexanox
Number analyzed (Participants) | 6
kg | -2.2 [-5.7 to -0.1]

ADVERSE EVENTS:
Time Frame: 16 weeks (12 weeks of treatment and 4 of followup)
Arm/Group | Amlexanox
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amlexanox (N=7)
elevated triglycerides (Blood and lymphatic system disorders) | 1
nausea (Gastrointestinal disorders) | 1
upper respiratory infection (Infections and infestations) | 2
restless legs (Nervous system disorders) | 1
polyuria (Renal and urinary disorders) | 1
Subcutaneous nodule at biopsy site (Skin and subcutaneous tissue disorders) | 1
breast abscess (Skin and subcutaneous tissue disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes